CLINICAL TRIAL: NCT03240809
Title: An Open-label, Single-dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Brodalumab in Pediatric Subjects (6 to < 18 Years Old) With Severe Plaque Psoriasis
Brief Title: An Open-label, Single-dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Brodalumab in Pediatric Subjects
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V01-BROA-401
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): (ages 12 to <18 years): 140 mg SC dose of brodalumab
  Interventions: Biological: Brodalumab
- Cohort 2 (Experimental): (ages 6 to <12 years): 70 mg SC dose of brodalumab
  Interventions: Biological: Brodalumab

INTERVENTIONS:
Biological: Brodalumab — 140 mg SC dose
  Arms: Cohort 1
Biological: Brodalumab — 70 mg SC dose
  Arms: Cohort 2

SUMMARY:
An Open-label, Single-dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Brodalumab in Pediatric Subjects

DETAILED DESCRIPTION:
An Open-label, Single-dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Brodalumab in Pediatric Subjects (6 to < 18 Years Old) With Severe Plaque Psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Subject's parent(s) or legally acceptable representative has provided informed consent, using an Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved Informed Consent Form (ICF), when the subject is legally too young to provide informed consent and the subject has provided written assent based on local regulations and/or guidelines prior to any study-specific activities/procedures being initiated, or when the subject has any kind of condition that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent.
2. Males and females ages 6 to <18 years of age, inclusive, at the time of screening
3. Subjects must have up-to-date immunizations according to the relevant local country guideline. Subjects must not be scheduled to be vaccinated while on study.
4. Female subjects of childbearing potential must have a negative serum pregnancy test at screening and a negative serum or urine pregnancy test at Baseline (Day 1). A female of childbearing potential is defined as a female who is fertile, following menarche.

Exclusion Criteria:

1. Received conventional systemic therapies or phototherapy for treatment of psoriasis within the last 4 weeks. Topical corticosteroids are allowed.
2. Female subjects who have reached puberty and are sexually active and are unwilling to use acceptable methods of effective birth control for the duration of the study and continuing for 5 weeks after receiving the dose of study drug. Acceptable methods of effective birth control include sexual abstinence (males and females); double barrier method (male condom with spermicide in combination with one female barrier method [diaphragm, cervical cap, or contraceptive sponge)]; or hormonal birth control; or intra-uterine device.
3. Female subjects who are lactating/breastfeeding or who plan to breastfeed while on study through 5 weeks after receiving the dose of study drug.
4. Female subjects with a positive pregnancy test.
5. Female subjects who are pregnant or planning to become pregnant while on study through 5 weeks after receiving the dose of study drug.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
maximum observed concentration (Cmax) | 29 Days
  maximum (or peak) serum concentration that drug achieves in the body after drug has been administrated and prior to the administration of a second dose

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Bhatt, Study Director — Bausch Health
Locations (5):
- United States (5):
  - Bausch Site 003, San Diego, California
  - Bausch Site 002, Miami, Florida
  - Bausch Site 004, Miami, Florida
  - Bausch Site 005, Henderson, Nevada
  - Bausch Site 001, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Undecided